CLINICAL TRIAL: NCT07322835
Title: Efficacy and Safety of Reperfusion Therapy for Minor Ischemic Stroke in China: A Multicenter Prospective Cohort Study
Brief Title: Efficacy and Safety of Reperfusion Therapy for Minor Ischemic Stroke in China
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinsheng Zeng, MD, PhD, Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: RERISE
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Minor Ischemic Stroke
Keywords: minor ischemic stroke; reperfusion therapy; intravenous thrombolysis; endovascular therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reperfusion therapy cohort: intravenous thrombolysis ± endovascular therapy, endovascular therapy alone
- Standard of care cohort: Recommended by guidelines for secondary stroke prevention, e.g. dual/mono antiplatelet, antihypertensive or lipid-lowing therapy, et al

SUMMARY:
Acute ischemic stroke is the most common type of stroke in China, accounting for 69.6% -72.8% of new strokes. In recent years, the proportion of mild stroke (NIHSS ≤ 5 points) has gradually increased, exceeding 50%, and the recurrence rate of stroke within one year is 13.2%, with a mortality rate of 6.3%, and 4% -10% may experience early deterioration of neurological function within 72 hours. At present, the main treatment for mild ischemic stroke is antiplatelet aggregation or anticoagulation drugs, but there are still 10% -20% of patients with residual neurological disability. There is still controversy over whether acute reperfusion therapy (including intravenous thrombolysis and endovascular intervention therapy) can improve the prognosis of such patients. In addition, it has been confirmed that beyond the time window thrombolysis is effective for selected ischemic stroke patients, but it is urgent to clarify whether mild ischemic stroke patients can benefit from receiving beyond the time window thrombolysis. Due to the limited evidence and inconsistent conclusions on the efficacy and safety of reperfusion therapy in patients with mild stroke, it is urgent to have a deeper understanding of the current status of reperfusion therapy for mild ischemic stroke in China based on real clinical data, and systematically compare the efficacy and safety of reperfusion therapy (including intravenous thrombolysis and endovascular intervention therapy) with standard drug therapy for this type of patient. This project plans to conduct a nationwide multicenter prospective cohort study to evaluate the differences in excellent neurological function prognosis (mRS ≤ 1) and symptomatic intracranial hemorrhage rate among patients with mild ischemic stroke who receive reperfusion therapy (intravenous thrombolysis ± endovascular intervention therapy) compared to standard drug therapy at 90 days, in order to guide accurate clinical decision-making. The research results have significant implications for improving the prognosis of patients with mild ischemic stroke, and will also lay an important foundation for future large-scale randomized controlled studies to explore the optimal treatment strategies for mild stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 year
2. Pre-stroke mRS ≤1
3. Diagnosis of ischemic stroke, confirmed by imaging (CT or MRI)
4. Stroke onset or last seen well (LSW) to visit ≤ 24h
5. NIHSS ≤ 5
6. Receive standard medication or IVT (TNK or rtPA) ± EVT, or EVT alone; for IVT beyond standard time window, initiation of treatment must occur within 4.5-24h of last seen well and ASPECTs≥7 or Perfusion lesion-ischemic core mismatch (ischemic core volume <70mL, mismatch rate >1.2, mismatch volume >10mL or mismatch between the presence of an abnormal signal on DWI and no visible signal change on FLAIR)
7. Patients or their eligible surrogates provided informed consent

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Patients who already received reperfusion therapy for the current stroke before arriving at the hospital
3. Participation in another interventional clinical trial that could interfere with the outcomes of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with minor ischemic stroke (NIHSS ≤ 5) within 24h from onset
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of modified Rankin scale score 0-1 | Day 90
  Modified Rankin Scale score ranges from 0 to 6, and lower score means better functional independence.

SECONDARY OUTCOMES:
Proportion of Modified Rankin Scale score 0-2 | Day 90
  Modified Rankin Scale score ranges from 0 to 6, and lower score means better functional independence.
Proportion of Modified Rankin Scale score 0-3 | Day 90
  Modified Rankin Scale score ranges from 0 to 6, and lower score means better functional independence.
Ordinal Modified Rankin Scale score | Day 90
  Modified Rankin Scale score ranges from 0 to 6, and lower score means better functional independence.
Change from baseline in National Institutes of Health Stroke Scale | Hour 24
  National Institutes of Health Stroke Scale ranges from 0 to 42, and higher score indicates more severe neurologic deficits.
Change from baseline in National Institutes of Health Stroke Scale | Hour 72
  National Institutes of Health Stroke Scale ranges from 0 to 42, and higher score indicates more severe neurologic deficits.
National Institutes of Health Stroke Scale | Day 7 or discharge (whichever comes first)
  National Institutes of Health Stroke Scale ranges from 0 to 42, and higher score indicates more severe neurologic deficits.
Barthel Index score | Day 90
  Barthel Index ranges from 0 to 100, and higher score means more functional independence.
Proportion of patients with door-to-needle time < 60 minutes | immediately after the intervention

OTHER OUTCOMES:
Proportion of symptomatic intracerebral hemorrhage (ECASS III) | Day 7 or discharge
Proportion of moderate or severe systemic bleeding (The GUSTO criteria) | Day 7 or discharge
Mortality | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Jinsheng Zeng, MD, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided